CLINICAL TRIAL: NCT04444011
Title: A Single-center, Randomized, Open-label, Crossover Study to Evaluate the Pharmacokinetic Drug-drug Interaction of the Quadruple Therapy With Anaprazole/Amoxicilin/Clarithromycin/Bismuth in Healthy Chinese Male Subjects
Brief Title: Pharmacokinetic Interactions of Quadruple Therapy With Anaprazole/Amoxicilin/Clarithromycin/Bismuth
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sihuan Pharmaceutical Holdings Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3571-DDI-1006
Record Dates: First submitted 2020-05-15; First posted 2020-06-23 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-03

CONDITIONS: Healthy Male Volunteers
MeSH Terms: interventions — Amoxicillin; Clarithromycin; Bismuth

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Anaprazole Sodium enteric-coated tablet (Experimental): Administered orally twice daily (e.g., 8am,8pm) for 5 consecutive days in 1 of 4 treatment periods of cohort 1 ( only once on the morning of D5 of treatment periods), one tablet each time.
  Interventions: Drug: Anaprazole Sodium
- Amoxicillin capsules (Experimental): "Administered orally twice daily (e.g., 8am,8pm) for 5 consecutive days in 1 of 4 treatment periods of cohort 1 ( only once on the morning of D5 of treatment periods), 2 capsules each time.
  Interventions: Drug: Amoxicillin
- Clarithromycin tablet (Experimental): "Administered orally twice daily (e.g., 8am,8pm) for 5 consecutive days in 1 of 4 treatment periods of cohort 1 ( only once on the morning of D5 of treatment periods), 2 tablets each time.
  Interventions: Drug: Clarithromycin
- Anaprazole + Amoxicillin +Clarithromycin (Experimental): "Cohort 1: Administered orally twice daily (e.g., 8am,8pm) for 5 consecutive days in 1 of 4 treatment periods ( only once on the morning of D5 of treatment periods).
  Cohort 2: Administered orally on an empty stomach once on the morning of D1 of treatment periods
  Interventions: Drug: Anaprazole Sodium; Drug: Amoxicillin; Drug: Clarithromycin
- Anaprazole + Amoxicillin +Clarithromycin+Bismuth (Experimental): Administered orally on an empty stomach once on the morning of D1 of treatment periods in cohort 2
  Interventions: Drug: Anaprazole Sodium; Drug: Amoxicillin; Drug: Clarithromycin; Drug: Bismuth

INTERVENTIONS:
Drug: Anaprazole Sodium — Anaprazole Sodium isthePPI inhibitor
  Arms: Anaprazole + Amoxicillin +Clarithromycin; Anaprazole + Amoxicillin +Clarithromycin+Bismuth; Anaprazole Sodium enteric-coated tablet
Drug: Amoxicillin — antibiotic
  Arms: Amoxicillin capsules; Anaprazole + Amoxicillin +Clarithromycin; Anaprazole + Amoxicillin +Clarithromycin+Bismuth
Drug: Clarithromycin — antibiotic
  Arms: Anaprazole + Amoxicillin +Clarithromycin; Anaprazole + Amoxicillin +Clarithromycin+Bismuth; Clarithromycin tablet
Drug: Bismuth — Bismuth is to protect the gastric mucosa
  Arms: Anaprazole + Amoxicillin +Clarithromycin+Bismuth

SUMMARY:
A single-center, randomized, open-label, crossover study to evaluate the pharmacokinetic drug-drug interaction and safety of the quadruple therapy with Anaprazole 20mg/Amoxicilin 1000mg/Clarithromycin 500mg/Bismuth Potassium Citrate 0.6g in healthy Chinese male subjects.

DETAILED DESCRIPTION:
The study composed of 2 cohorts, using a 4*4 or 2*2 crossover design in cohort 1 and 2, respectively. 4 rotating treatment sequences in cohort 1, each treatment sequence comprised 4 treatment periods, separated by a washout period of 9 days; 2 rotating treatment sequences in cohort 2, each treatment sequence comprised 2 treatment periods, separated by a washout period of 9 days

ELIGIBILITY:
Inclusion Criteria:

* 1.The subject is capable of understanding and complying with protocol requirements, and signed and dated a written informed consent form voluntarily
* 2.The subject is a Chinese adult male, aged 18 to 35 years, inclusive.
* 3.The subject is a H. pylori-negative via UBT.
* 4.The subject weighed at least 50.0 kg and had a body mass index (BMI) between 19.0 kg/m^2 and 26.0 kg/m^2, inclusive.
* 5.Has clinical laboratory evaluations, vital signs and ECG testing within the reference range, and medical history and physicial examination results are normal. Participants with evaluations outside the reference range that are deemed not clinically significant by the investigator may be included at investigator discretion
* 6.The subject with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for 3 months after last dose.
* 7.The subjects have a good lifestyle and can keep good communication with the investigators and comply with the requirements of clinical trial

Exclusion Criteria:

* 1.Has clinical significant drug allergy or allergic disease history(Such as asthma, urticaria, eczema dermatitis, etc), or has hypersensitivity or allergy to investigatory drugs or related supplements；
* 2.Has clinical significant ECG abnormal history or family history of long QT syndrome(Grandparents, parents and siblings)
* 3.Any disease or medical history that may significantly affect the absorption, distribution, metabolism, and excretion of drugs, or any condition that may pose a hazard to the subject. Such as:

  * Inflammatory bowel disease, gastric ulcer, duodenal ulcer, gastrointestinal / rectal bleeding, persistent nausea, or other clinically significant gastrointestinal abnormalities;
  * Has suffered from gastrointestinal diseases or complications that may affect the absorption of drugs (ie: malabsorption, gastroesophageal reflux, peptic ulcer, erosive esophagitis, frequent heartburn) within 6 months before screening or had history of gastrointestinal surgery (for example: gastrectomy, gastrointestinal anastomosis, intestinal resection, gastric bypass, gastric segmentation or gastric banding, cholecystectomy, except for appendicitis surgery and proctectomy);
  * Evidence of liver disease or clinically impaired liver function at the time of screening (eg AST, ALT or total bilirubin> 1.5 times ULN);
  * A history or evidence of nephropathy or renal insufficiency at the time of screening, showing clinically significant abnormality of creatinine or abnormal urine composition (such as proteinuria, creatinine> 176.8 umol / L, etc.)
  * Has difficulty swallowing oral preparations.
* 4.Thyroid stimulating hormone (TSH)> ULN; or serum free triiodothyronine (FT3)> ULN; or serum free thyroxine (FT4)> ULN at the time of screening;
* 5. Frequent smokers and alcoholics within 3 months before screening (smoke more than 5 cigarettes / day, drink more than 21 units of alcohol per week, 1 unit = 360 mL beer or 45 mL liquor or 150 mL wine), or can't stop using any tobacco products, and alcohol intake during the study period ; or those who have a positive alcohol breath test before enrollment;
* 6. Has received any investigational compound (including post-marketing investigational drugs) or participated in clinical trials of any drugs /devices within 3 months before screening;
* 7. A history of drug abuse within 12 months before screening or a positive urine test result at screening;
* 8. Has used any prescription drugs, non-prescription drugs (including chemical drugs, vitamin drugs, Chinese herbal medicines, etc.) within 4 weeks before administration of investigational drugs;
* 9. Has taken foods that affect CYP3A4 (such as grapefruit or beverages containing grapefruit) within 2 weeks before administration of investigational drugs;
* 10. Human immunodeficiency virus antibody, hepatitis B surface antigen, hepatitis C antibody, and Treponema pallidum specific antibody test results were positive at screening;
* 11. Has difficulty in venous blood collection or halo acupuncture;
* 12.Blood donation / blood loss ≥200 mL within 1 month, or ≥400 mL within 3 months before screening; or has blood donation plan during the period of medication of investigational drugs and within 3 months after drug withdrawal;
* 13. Has special dietary requirements and cannot follow the unified dietary arrangements;
* 14. Any conditions in which considered by investigator not be appropriate to participate in this trial.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-10-15 (Estimated)

PRIMARY OUTCOMES:
Cohort 1: Css,max of anaprazole (parent drug, KBP-3571) and its enantiomer（KBP-3570）and its major metabolites (KBP-1123 and KBP-1144), Unchanged amoxicillin, Unchanged clarithromycin and its metabolite (14-hydroxyclarithromycin) | Hour 0.5 pre-dose and 0.5，1，1.5，2，2.5，3，3.5，4，4.5，5，6，7，8，10，12，24 hours post-dose of Day 5，Day 19，Day 33，Day 47
  Css,max is the peak plasma concentration at steady state
Cohort 1: AUC of anaprazole (parent drug, KBP-3571) and its enantiomer（KBP-3570）and its major metabolites (KBP-1123 and KBP-1144), Unchanged amoxicillin, Unchanged clarithromycin and its metabolite (14-hydroxyclarithromycin) | Hour 0.5 pre-dose and 0.5，1，1.5，2，2.5，3，3.5，4，4.5，5，6，7，8，10，12，24 hours post-dose of Day 5，Day 19，Day 33，Day 47
  AUC is area under the plasma concentration-time curve
Cohort 2: Cmax of anaprazole (parent drug, KBP-3571) and its enantiomer（KBP-3570）and its major metabolites (KBP-1123 and KBP-1144), Unchanged amoxicillin, Unchanged clarithromycin and its metabolite (14-hydroxyclarithromycin) | Hour 0.5 pre-dose and 0.5，1，1.5，2，2.5，3，3.5，4，4.5，5，6，7，8，10，12，24 hours post-dose of Day 1，Day 11
  Cmax is the peak plasma concentration
Cohort 2: AUC of anaprazole (parent drug, KBP-3571) and its enantiomer（KBP-3570）and its major metabolites (KBP-1123 and KBP-1144), Unchanged amoxicillin, Unchanged clarithromycin and its metabolite (14-hydroxyclarithromycin) | Hour 0.5 pre-dose and 0.5，1，1.5，2，2.5，3，3.5，4，4.5，5，6，7，8，10，12，24 hours post-dose of Day 1，Day 11
  AUC is area under the plasma concentration-time curve

SECONDARY OUTCOMES:
Number of subjects with adverse events and serious adverse events as assessed by CTCAE v5.0 | From signing informed consent to study completion. 56 days minimum, 68 days maximum(Cohort 1); 30 days minimum, 32 days maximum(Cohort 2)
  All adverse events will be monitored in each subject